CLINICAL TRIAL: NCT03076957
Title: A Phase 1/2a Study to Assess the Safety and Efficacy of CKD-516 Tab. in Combination With Irinotecan Inj. in Patients With Previously Treated Advanced Colorectal Cancer
Brief Title: A Phase 1/2a Study to Assess the Safety and Efficacy of CKD-516 Tab. in Combination With Irinotecan Inj.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127CRC16009
Record Dates: First submitted 2016-12-22; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(4-(3-(1H-1,2,4-triazol-1-yl)-4-(3,4,5-trimethoxybenzoyl)phenyl)thiazol-2-yl)-2-amino-3-methylbutanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treat Regimen (Experimental): CKD-516(investigational Drug) Irinotecan
  Interventions: Drug: CKD-516 Tablet

INTERVENTIONS:
Drug: CKD-516 Tablet — CKD-516 PO for 5 consecutive days and 2 days off in Combination with Irinotecan inj.
  Other Names: CKD-516

SUMMARY:
The purpose of this open-label, dose-escalation phase I trial is to evaluate the safety, tolerability and pharmacokinetic profiles and to assess the efficacy of CKD-516 Tablet in Combination with Irinotecan inj. in Patients with Previously Treated Advanced Colorectal Cancer

DETAILED DESCRIPTION:
CKD-516 tab. in combination with Irinotecan inj.(1cycle=14days)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 19 years or older
2. Patients who failed existing anti-cancer therapies
3. ECOG performance status ≤ 1
4. Life expectancy of ≥ 12 weeks
5. Adequate hematological, hepatic and renal functions:
6. Patients who give written informed consent voluntarily

Exclusion Criteria:

1. Prior systemic chemo-, radiochemo-, radio-, immuno-, hormonal and/or biological therapy within 2 weeks before study participation (in case of nitrosoureas and/or mitomycin, within 6 weeks before study participation)
2. Patients who received major surgery within 4 weeks before study participation (in case of VATS and/or ONC surgery, within 2 weeks before study participation)
3. Symptomatic CNS metastases (patients with radiologically and neurologically stable metastases and being off corticosteroids for at least 4 weeks are able to participate in this trial.)
4. NYHA class III or IV heart failure, uncontrolled hypertension (SBP/DBP > 140/90 mm Hg), other clinically significant cardiovascular abnormalities at investigator's discretion (e.g., LVEF < 50%, clinically significant cardiac wall abnormalities or cardiac muscle damages)
5. Acute coronary syndrome (unstable angina or myocardial infarction) within 6 months
6. Uncontrolled arrhythmia
7. Significant cerebrovascular diseases including stroke within 6 months
8. Significant vascular diseases including aortic aneurysm requiring treatment or peripheral arterial diseases
9. Patients with known active hepatitis, HIV infection, or other uncontrolled infectious disease
10. Patients who cannot receive IP by mouth and have a history of clinically significant gastrointestinal disorders which can impede administration, transit or absorption of the IP
11. A history of severe drug hypersensitivity or hypersensitivity to analogs of the IP
12. Pregnancy or breast-feeding
13. Women of childbearing potential (WOCBP) or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 3 months after the end of treatment
14. Patients who received other investigational products or used other investigational devices within 3 weeks before participation
15. Patients who cannot participate in this trial by investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | Up to 14 days(for 1st cycle)

SECONDARY OUTCOMES:
Pharmacokinetics(Cmax) | 1st Cycle Day1: up to 24hr
Number of participants with toxicity as assessed by CTCAE v4.03 through study completion, an average of 1 year | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tae won KIM, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jeong H, Hong YS, Kim JE, Lim HS, Ahn JB, Shin SJ, Park YS, Kim ST, Han SW, Kim TY, Kim TW. A phase 1 dose-escalation and dose-expansion study to assess the safety and efficacy of CKD-516, a novel vascular disrupting agent, in combination with Irinotecan in patients with previously treated metastatic colorectal cancer. Invest New Drugs. 2021 Oct;39(5):1335-1347. doi: 10.1007/s10637-021-01110-9. Epub 2021 Apr 7. PMID 33829355